CLINICAL TRIAL: NCT07192809
Title: Chronic Non-Specific Low Back Pain: Investigating the Effectiveness of a Dual-Task Program as an Attention Distraction Strategy
Brief Title: The Effect of Attention Distraction on the Adherence to Exercise, in Chronic Low Back Pain Patients.
Acronym: PAINLESS
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Thessaly (Other)
Responsible Party: Principal Investigator, Savvas Spanos, Supervising Professor Dr Savvas Spanos, University of Thessaly
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 20787/25/TFSKTH - 09/07/2025
Record Dates: First submitted 2025-07-13; First posted 2025-09-25 (Actual); Last update posted 2025-09-25 (Actual); Status verified 2025-09

CONDITIONS: Chronic Low Back Pain (CLBP); Distraction Methods; Adherence to Care
Keywords: chronic low back pain; adherence; distraction; divided attention; chronic non specific low back pain

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Distraction Group (Experimental): Experimental Group: Standard exercise program with Attention Distraction Application (AD-APP)
  Participants in this group will:
  * will be familiarized with the exercises on a separete day prior to testing.
  * Perform exercises while using an application designed to distract attention in order to achieve a cognitive-motor dual task (exercise task and cognitive task).
  * Follow the program for 8 weeks, attending non-supervised sessions per week. Every two weeks , there will be a progression that will be achieved by increasing the level of difficulty of each exercise.
  * Adherence to the exercise program will be tracked through digital monitoring within the application.
  * Stratified into IPAQ categories (low, moderate, high physical activity).
  Participants will be given special equipment including an elastic tubing load Thera BandTM (Akron, Ohio, USA).
  Interventions: Other: Stabilisation exercise, resistance exercise and distraction task
- Control Group (Active Comparator): Control Group: Standard exercise program without Attention Distraction Application (AD-APP)
  Participants in this group will:
  * will be familiarized with the exercises on a separete day prior to testing.
  * Perform the same exercises without attention distraction in order to achieve a single task (exercise task).
  * Follow the program for 8 weeks, attending non-supervised sessions per week.
  * Adherence to the exercise program will be tracked through EARS-GR.
  * Stratified into IPAQ categories (low, moderate, high physical activity).
  Participants will be given special equipment including an elastic tubing load Thera BandTM (Akron, Ohio, USA).
  Interventions: Other: stabilisation exercise and resistance exercises

INTERVENTIONS:
Other: Stabilisation exercise, resistance exercise and distraction task — The 8-week exercise intervention consists of 25 minutes non supervised training while distracting their attention with a knowledge based application
  Arms: Distraction Group
Other: stabilisation exercise and resistance exercises — The 8-week exercise intervention consists of 25 minutes non supervised training without distracting their attention with a knowledge based application
  Arms: Control Group

SUMMARY:
This randomized controlled trial aims to investigate whether the use of an attention distraction application during exercise increases patient adherence to exercise programs in chronic non-specific low back pain (CNSLBP). In addition, the study will examine whether higher adherence to exercise leads to improved outcomes in pain levels, functional capacity, kinesiophobia, quality of life, central sensitization, and pain catastrophizing.

DETAILED DESCRIPTION:
Participants will be stratified based on their level of physical activity according to the International Physical Activity Questionnaire (IPAQ) into:

* Low physical activity
* Moderate physical activity
* High physical activity

They will then be randomly assigned to one of two groups: (1) an experimental group using the attention distraction application during the standard exercise program and (2) a control group following the same standard exercise program without distraction. The intervention will last for 8 weeks, with participants attending three non-supervised sessions per week (total: 24 training sessions). Each session will last approximately 25-30 minutes. Adherence to the exercise program will be monitored through the EARS questionnaire and the distraction application (The total score ranges from 0 to 24, where a higher score reflects better adherence).

The intervention group sessions consist of 5 minute submaximal warm-up followed by 25 minutes of stabilisation and resistance training with exercises focused on strength and stabilisation while using the distraction application. The training will consist of two parts: warming-up and the resistance and stabilisation program. The resistance program will consist of 4 exercises: knee flexion, abdominal crunches, prone superman and leg extension. Each exercise will be performed for 3 sets of 10 repetitions with a rest of 30 sec corresponding to every set , and 1 minute between each exercise. The stabilisation program will consist of 3 exercises: bridge, plank and side plank. Each exercise will be performed for 3 sets of 1 repetition (maximum time) with a rest of 30 sec corresponding to every set and 1 minute between each exercise. Four levels of difficulty will be given for each exercise to allow for progression. Every 2 weeks, there will be a progression that will be achieved by increasing the resistance band tension, by changing the base of support or my modifying the length of resistance level arm.

In the control group they will perform the same exercises without the distraction-based application.

The exercise intensity will be monitored by the researcher, as determined by the patient's ability to complete three sets of 8-12 repetitions for a given exercise and a CR10scale. The progression will be in line with guidelines provided by the American College of Sports Medicine.

Adherence to the program for both groups will be assessed by the Exercise Adherence Rating Scale (EARS - GR).

ELIGIBILITY:
Inclusion Criteria:

* Age > 18 years
* Chronic non-specific low back pain (≥3 months)
* No physical therapy or structured exercise program in the last 3 months
* Willingness to use the attention distraction application (for the AD-APP group)
* Completion of the International Physical Activity Questionnaire (IPAQ)

Exclusion Criteria:

* History of spinal surgery
* Neurological conditions affecting movement
* Regular use of pain relief medication within the past two weeks
* Pregnancy
* Severe psychological disorders that may affect compliance

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2025-09-20 (Estimated); Primary Completion 2026-01-31 (Estimated); Study Completion 2026-01-31 (Estimated)

PRIMARY OUTCOMES:
Adherence to exercise | Baseline, Week 8, and follow-up (6 months).
  Exercise Adherence Rating Scale in Greek (EARS-GR).
  The Exercise Adherence Rating Scale (EARS) is a questionnaire used to assess how well individuals adhere to prescribed exercise programs. It utilizes a 5-point Likert scale for each item, with higher scores indicating better adherence. The total score ranges from 0 to 24, with higher scores representing greater adherence.
Adherence to exercise | During the 6 month intervention period.
  Measured through app recorded metrics, including number of sessions (number)
Adherence to exercise | During the 6 month intervention period.
  Measured through app recorded metrics, including duration per session (minutes)
Adherence to exercise | During the 6 month intervention period
  Measured through app recorded metrics including frequency of use per week (minutes)
Adherence to exercise | During the 6 month intervention period
  Measured through app recorded metrics, including number of questions answered
Adherence to exercise | During the 6 month intervention period
  Measured through app recorded metrics, including total active time (minutes).

SECONDARY OUTCOMES:
Pain Intensity | Baseline, Week 8, and follow-up (6 months).
  Numeric Pain Rating Scale (NPRS).
  The Numeric Pain Rating Scale (NPRS) is a widely used tool for assessing pain intensity, typically ranging from 0 to 10. In this scale, 0 represents no pain, and 10 represents the worst pain imaginable. Patients are asked to verbally select a number that best reflects their pain level.
Anxiety, Stress, and Depression | Baseline, Week 8, and follow-up (6 months).
  Depression, Anxiety, and Stress Scale (DASS-21).
  The Depression Anxiety Stress Scales 21 (DASS-21) is scored by summing the responses to each of the three subscales: Depression, Anxiety, and Stress. Each subscale contains 7 items, and each item is scored on a scale of 0 to 3. The raw scores for each subscale are then multiplied by 2 to get the final score for each domain, which can range from 0 to 42.
Functionality | Baseline, Week 8, and follow-up (6 months).
  Oswestry Disability Index (ODI).
  The Oswestry Disability Index (ODI) is scored out of a total of 50 points, with each of the 10 sections having a maximum score of 5. To calculate the ODI score, sum the scores for each section, divide by the total possible score (50), and multiply by 100 to express it as a percentage.
Pain Catastrophizing | Baseline, Week 8, and follow-up (6 months).
  Pain Catastrophizing Scale (PCS).
  The Pain Catastrophizing Scale (PCS) is a 13-item questionnaire used to assess pain catastrophizing, with higher scores indicating greater levels of catastrophizing. Scores range from 0 to 52, and a score above 30 is considered clinically significant. The PCS also has three subscales: rumination, magnification, and helplessness.
Central Sensitization | Baseline, Week 8, and follow-up (6 months).
  Central Sensitization Inventory (CSI).
  The CSI, or Central Sensitization Inventory, is a questionnaire used to assess the severity of Central Sensitization Syndrome (CSS). It consists of 25 questions (Part A) scored on a 5-point Likert scale, with higher scores indicating more severe symptoms. Part B is not used for scoring but provides additional clinical information. The total score ranges from 0 to 100, with different ranges corresponding to different severity levels: subclinical (0-29), mild (30-39), moderate (40-49), severe (50-59), and extreme (60-100).
Kinesiophobia | Baseline, Week 8, and follow-up (6 months)
  Tampa Scale of Kinesiophobia (TSK).
  The Tampa Scale for Kinesiophobia (TSK) is a questionnaire used to assess fear of movement or re-injury, often related to chronic pain conditions. Scoring involves summing the responses to each item, with higher scores indicating greater kinesiophobia. The original TSK has 17 items, while a shorter version, TSK-11, has 11 items. The TSK-11 is more commonly used due to its reduced administration time and similar psychometric properties.
Individual's health-related quality of life | Baseline, Week 8, and follow-up (6 months)
  12-Item Short Form Survey (SF-12)
  The SF-12v2 scoring provides a Physical Component Summary (PCS) and a Mental Component Summary (MCS) score, both with a mean of 50 and a standard deviation of 10 in the US general population. Higher scores indicate better health on both scales. These scores are derived from the 12 individual items, which are scored and then transformed using regression weights to generate the PCS and MCS scores.
Effect of Physical Activity Level | Analyzed post-intervention based on IPAQ stratification
  International Physical Activity Questionnaire (IPAQ).The patients will be categorized based on their level of physical activity, and accordingly, they will be assigned different exercise programs. Depending on their activity level, patients will perform exercises with a corresponding number of repetitions, weekly frequency, and intensity.
  The International Physical Activity Questionnaire (IPAQ) scoring involves calculating Metabolic Equivalent of Task (MET) minutes per week to assess physical activity levels. The IPAQ scoring protocol provides guidelines for data processing and analysis, including recommendations for data cleaning. There are two main ways to express the results: as a continuous variable (MET-minutes per week) or categorized into low, moderate, or high activity levels. Investigate whether baseline physical activity level influences outcomes
Work Productivity | Baseline, Week 8, and follow-up (6 months)
  Work Productivity and Activity Impairment Questionnaire - General Health (WPAI-GH Greek).
  The Work Productivity and Activity Impairment Questionnaire - General Health (WPAI:GH) is a tool used to assess the impact of general health problems on work and daily activities over the past seven days. It consists of six questions that evaluate employment status, hours missed from work due to health problems, hours missed for other reasons, hours actually worked, and the degree to which health problems affected productivity while working and during regular daily activities. The last two questions are scored on a scale of 0 to 10, with 0 indicating no effect and 10 indicating complete impairment.
Lumbar Mobility | Baseline, Week 8, and follow-up (6 months).
  Modified-Modified Schober Test.
  The modified-modified Schober test (MMST) is a clinical assessment used to measure lumbar flexion range of motion. It involves marking two points on the back and measuring the distance between them while the patient bends forward, helping to quantify and track lumbar spine flexibility.
Muscle Endurance | Baseline, Week 8, and follow-up (6 months).
  Modified Biering-Sorensen Test.
  It shows that maintaining the Biering-Sorenson position for less than 176 seconds, predicts low back pain within the next year and greater than 198 seconds predicts absence of low back pain. It also reported that Biering-Sorenson test does not have a ceiling effect.
Gait Analysis | Baseline, Week 8, and follow-up (6 months).
  Kinovea software for gait assessment.
  The following parameter will be assessed using Kinovea software: step length (cm).
Gait Analysis | Baseline, week 8 and follow - up (6 months)
  Kinovea software for gait assessment. The following parameter will be assessed using Kinovea software: stride length (cm).
Gait Analysis | Baseline, Week 8 and follow-up (6 months).
  Kinovea software for gait assessment. The following parameter will be assessed using Kinovea software: knee range of motion (degrees).
Gait analysis | Baseline, week 8 and follow-up (6 months)
  Kinovea software for gait assessment. The following parameter will be assessed using Kinovea software: ankle angle (degrees).
Gait analysis | Baseline, week 8 and follow-up (6 months)
  Kinovea software for gait assessment. The following parameter will be assessed using Kinovea software: knee angle (degrees).
Gait analysis | Baseline, Week 8 and follow- up (6 months)
  Kinovea software for gait assessment. The following parameter will be assessed using Kinovea software: pelvic tilt (degrees).
Gait analysis | Baseline, Week 8 and follow-up (6 months)
  Kinovea software for gait assessment. The following parameter will be assessed using Kinovea software: base of support (cm).

CONTACTS AND LOCATIONS:
Locations (1):
- University of Thessaly, Lamia, Central Greece, Greece